CLINICAL TRIAL: NCT00336050
Title: Fresno Asthmatic Children's Environment Study
Brief Title: Effect of Air Pollution on Long-Term Asthma Severity and Lung Function in Children
Acronym: FACES
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Mickey Leland National Urban Air Toxics Research Center (Other)
Responsible Party: Ira B. Tager, MD, MPH, School of Public Health, University of California, Berkeley
Other Study IDs: 1341; R01HL081521-01A1 (NIH)
Record Dates: First submitted 2006-06-09; First posted 2006-06-12 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2009-02

CONDITIONS: Asthma
Keywords: Air Pollution; Pulmonary Function
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Password-protected database and storage facility that is part of the UCB SPH biorepository
Oversight: Data Monitoring Committee: No

SUMMARY:
Asthma can be caused by many factors, including mold, pollen, and other airborne pollutants. The purpose of this study is to evaluate the effect that air pollution has on the long-term severity of asthma symptoms and lung function in children.

DETAILED DESCRIPTION:
Asthma prevalence has steadily increased in the United States since the early 1980's; currently more than 20 million people are diagnosed with asthma, including 9 million children. Asthma can be caused by many factors, including pollen, dust, tobacco smoke, and other allergens. Research has shown that even short-term increases in daily levels of air pollution can trigger an increase in asthma symptoms in some individuals. More research is needed to determine how short-term increases in air pollution affect the severity of asthma later in life. The Environmental Protection Agency (EPA) has constructed research monitoring stations, known as Supersites, to advance the understanding of the effect of airborne pollutants on the health of individuals. Data collected from the Supersites provide important information regarding air pollution and air quality levels. This study will use air pollution measurements obtained from the Fresno, California Supersite to monitor participants' exposure to air pollution. The purpose of the study is to determine if children who experience a worsening of asthma symptoms due to an increase in air pollution have greater long-term asthma severity and decreased lung function compared to children who do not experience a worsening of symptoms when exposed to air pollution.

This study will enroll children with asthma who live within 20 kilometers of the EPA Supersite in Fresno, California. Participants will have study visits twice a year for up to 2 ½ years. At study entry, participants will undergo a skin prick allergy test and complete a dietary questionnaire. At each study visit, a respiratory illness questionnaire will be completed, and participants will undergo spirometry tests to measure lung function. In addition to the twice yearly visits, participants will take part in three 14-day sessions each year, during which daily diaries will be completed and spirometry will be performed twice a day. Study staff will gather detailed air pollution information from the Supersite, mobile monitoring trailers, and inside and outside the participants' homes.

Beginning in May 2006, participants will take part in only one study visit and two 14-day sessions each year. Air pollution measurements will be obtained from only the Supersite. To estimate daily exposure to air pollution, all participants will wear a global positioning system (GPS) device and complete daily activity diaries for 5 days during the school year. Fifty participants who have demonstrated compliance with study procedures will be selected to also wear the GPS devices for 5 days during the summer months.

The study completion date listed in this record was obtained from the "Completed Date" entered in the Query View Report System (QVR).

ELIGIBILITY:
Inclusion Criteria:

* Asthma, as diagnosed by study criteria, which includes experiencing asthma symptoms and/or use of specific asthma medications in the 12 months prior to study entry
* Resides within 20 kilometers of the EPA Supersite in Fresno, California
* Is not planning to move within 3 months of study entry

Exclusion Criteria:

* Current medical condition that would not allow individual to safely participate in the study

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Convenience sample of children ages 6-11 at intake with proven asthma. All live within a radius of 20 km from the EPA Super Site in Fresno, CA
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2000-11; Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Effect that air pollution has on the long-term severity of asthma symptoms and lung function in children | Measured during participants' study visits

CONTACTS AND LOCATIONS:
Overall Officials: Ira B. Tager, MD, MPH, Principal Investigator — School of Public Health, UC Berkeley